CLINICAL TRIAL: NCT00832299
Title: A Phase II Open- Labeled, Prospective Study to Determine the Efficacy of Pre- Operative Chemotherapy With Six Cycles of Modified FOLFOX 6 Followed by Total Mesorectal Excision (TME) Followed by an Additional Six Cycles of FOLFOX 6
Brief Title: Neo-Adjuvant FOLFOX for Rectal Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated for lack of enrollment
Sponsor: Beth Israel Medical Center (Other)
Collaborators: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-08; OX-08-006
Record Dates: First submitted 2009-01-27; First posted 2009-01-30 (Estimated); Results first posted 2013-04-22 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — Folfox protocol; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 6 cycles of FOLFOX pre and post TME (Experimental)
  Interventions: Drug: FOLFOX; Procedure: total mesorectal excision (TME)

INTERVENTIONS:
Drug: FOLFOX — 6 cycles of neo-adjuvant mFOLFOX6
  Other Names: oxaliplatin; leucovorin; 5-fluorouracil
Procedure: total mesorectal excision (TME) — TME will be done 4-6 weeks after 6 cycles of neo-adjuvant FOLFOX.
  Other Names: Total Mesorectal Excision

SUMMARY:
A Phase II open- labeled, prospective study to determine the efficacy of pre-operative chemotherapy with six cycles of modified FOLFOX 6 followed by total mesorectal excision (TME) followed by an additional six cycles of FOLFOX 6.

The objectives of this study are the following:

1. The primary endpoint of this trial is pathologic complete response (response rate).
2. Secondary endpoints will include observation of overall pathologic response rate, correlation of pathologic staging with pre-operative ultrasound and pelvic MRI staging, as well as observation of toxic side effects, patterns of disease relapse, disease-free survival outcomes and overall survival outcomes.

DETAILED DESCRIPTION:
Principal Investigator: Peter Kozuch, M.D.

Sites: BIMC/SLRHC

Introduction

A Phase II open- labeled, prospective study to determine the efficacy of pre-operative chemotherapy with six cycles of modified FOLFOX 6 followed by total mesorectal excision (TME) followed by an additional six cycles of FOLFOX 6.

The objectives of this study are the following:

1. The primary endpoint of this trial is pathologic complete response (response rate).
2. Secondary endpoints will include observation of overall pathologic response rate, correlation of pathologic staging with pre-operative ultrasound and pelvic MRI staging, as well as observation of toxic side effects, patterns of disease relapse, disease-free survival outcomes and overall survival outcomes.

Background Locally advanced rectal carcinoma continues to be a major oncologic problem in the United States. Several landmark studies have led to the current standard approach to the care of patients with stage II and III rectal cancer. In 1990 adjuvant 5- fluorouracil based chemoradiation became the accepted standard of care on the basis of two randomized trials. During the following two decades significant modifications were made to both the administration of chemoradiation therapy and surgery. First, continuous infusion 5-fluorouracil daily concurrent with radiation to was shown to be superior to bolus 5-fluorouracil for 3 consecutive days during weeks 1 and 5 of radiation. The overall rate of tumor relapse fell from 47% to 37%, and distant metastasis rate fell from 40% to 31%. Notably, local tumor recurrence was not significantly different between the two chemotherapy schedules. The improvement in relapse rate translated into a 4 year survival benefit, 70% versus 60%, favoring the protracted venous infusion of 5-fluorouracil (5-FU).

What is not known, however, is the relative contribution of radiation therapy to survival outcomes in the setting of chemotherapy programs for rectal cancer. Optimization of systemic therapy appears to have the most significant impact on survival outcomes. Firstly, patients may begin full systemic therapy with the regimen that has currently been identified as the most effective adjuvant treatment of stage III colon cancer. This relatively prompt initiation of 'full systemic dose' chemotherapy is in stark contrast to the typical paradigm of a 3-4 week interval between initial consultation and initiation of chemoradiation. Another theoretical advantage of this proposed trial lies in the fact that full systemic therapy is relatively uninterrupted. Therefore, the anticipated 6-8 week perioperative treatment free interval anticipated in this schema compares favorably with the typical 10-12 week perioperative treatment free interval with current standard of care neoadjuvant chemoradiation. Another important consideration favoring this chemotherapy is substantially less travel time/treatment time for patients and favorable toxicity profile given the elimination of daily neoadjuvant radiation.

Treatment Plan

Patients will be given:

* Modified FOLFOX6 will be given neoadjuvantly prior to resection for 3 months (6 cycles)
* Modified FOLFOX6 will be given adjuvantly within 6 weeks following resection for 3 months (6 cycles)

ELIGIBILITY:
Inclusion Criteria

1. Patients must consent to participate in the study and must have signed and dated an IRB-approved consent form conforming to federal and institutional guidelines
2. Patient must have histologically proven adenocarcinoma of the rectum with no distant metastases
3. Tumor stage must be T3N0M0, T1-3 N1M0 assessed by clinical exam, TRUS, MRI and CT. Pre-operative evidence of T4, N2 or distal lesions (0-6 cm from anal verge) should receive preoperative RT and not be offered this protocol. Any pT4, pN2 or CRM+ patients should be offered postoperative radiation
4. The proximal border of the tumor must be at or below 12 centimeters of the anal verge by proctoscopic examination
5. The distal border of the tumor must be at or above 6 cm from the anal verge on preoperative proctoscopy with the patient in the left lateral decubitus position
6. Patient must have had no prior chemotherapy or pelvic irradiation
7. Karnofsky performance status of 60 or greater; ECOG performance status 0-1
8. Patients should be age 18 years and older
9. Pretreatment absolute neutrophil count >= 1000/mm3 and platelets >= 100,000/mm3
10. Serum creatinine <= 1.5 x ULN; bilirubin <= 1.5 x ULN; ALT<= 2.5 x ULN

Exclusion Criteria

1. Patients can not be receiving any other investigational agents
2. Patients with known metastases will be excluded from the study
3. Patients with history of significant neuropathy or current symptoms of neuropathy
4. Patients with history of allergic reactions attributed to compounds of similar chemical or biologic composition to oxaliplatin or 5-FU or leucovorin
5. Patients with uncontrolled intercurrent illness not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
6. Pregnant women are excluded from this study because oxaliplatin and 5-FU/LV are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with oxaliplatin and 5-FU/LV, breastfeeding should be discontinued if the mother is treated with these agents
7. HIV positive patients
8. Patients with serious comorbid disease which prevents delivery of full treatment including psychiatric disorders and cardiopulmonary disease
9. No history within the past 5 years of a cancer diagnosis except for non-melanomatous skin cancers or in situ cervix carcinoma
10. Patients with clinically significant peripheral neuropathy at the time of start of treatment (defined in the NCI Common Terminology Criteria for Adverse Events Version 3[CTCAE v3.0] as grade 2 or greater neurosensory or neuromotor toxicity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kozuch, MD, Principal Investigator — Beth Israel Medical Center
Locations (2):
- United States (2):
  - Beth Israel Medical Center, New York, New York
  - St. Luke's Roosevelt Hospital Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the GI Oncology practice.
Groups:
- 6 Cycles of FOLFOX Pre and Post TME: total mesorectal excision (TME) : TME will be done 4-6 weeks after 6 cycles of neo-adjuvant FOLFOX.
  FOLFOX : 6 cycles of neo-adjuvant mFOLFOX6
Period: Overall Study
Arm/Group | 6 Cycles of FOLFOX Pre and Post TME
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 6 Cycles of FOLFOX Pre and Post TME
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response
Time Frame: 3-6 months
Population: Study terminated prior to data collection of time frame
Arm/Group | 6 Cycles of FOLFOX Pre and Post TME
Number analyzed (Participants) | 0

2. Secondary Outcome: Observation of Overall Pathologic Response Rate, Correlation of Pathologic Staging With Pre-op Ultrasound and Pelvic MRI Staging Observed Toxicities Patterns of Disease Relapse Disease-free Survival Overall Survival
Time Frame: 5 years
Population: Data not collected
Arm/Group | 6 Cycles of FOLFOX Pre and Post TME
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | 6 Cycles of FOLFOX Pre and Post TME
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes